CLINICAL TRIAL: NCT00526981
Title: Prone Position for Non-intubated Patients With Acute Respiratory Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Johan Petersson, MD, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007/733-31/1-4
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Prone position + all conventional treatment.
  Interventions: Other: Prone position
- Control (No Intervention): Conventional treatment

INTERVENTIONS:
Other: Prone position — Prone position during spontaneous breathing.
  Arms: Treatment

SUMMARY:
The study will test the hypothesis that the prone position can be used to reduce the need for intubation and mechanical ventilation in patients with acute respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* bilateral pulmonary infiltrates or unilateral infiltrates involving more than one lobe on CXR
* PaO2/FIO2 < 40 kPa
* RR > 25, or attending intensivist considering likelihood of intubation > 50%

Exclusion Criteria:

* unsuited for the prone position
* fulfilled inclusion criteria for more than 5 days (120 h)
* immunosuppression
* chronic lung disease
* decision of withdrawal or limitation of therapy
* pulmonary infiltrates of cardiac origin
* decreased GCS level
* PaCO2 > 10
* attending intensivist considering the patient unsuited for the prone position
* BMI > 33

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-09; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Need for intubation and mechanical ventilation | Duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Johan Petersson, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital Solna, Stockholm, Sweden